CLINICAL TRIAL: NCT02000414
Title: Pharmacokinetics Study of Intraperitoneal Administration of Daptomycin in Patients With Peritoneal Dialysis and Peritoneal Infection
Brief Title: Pharmacokinetics Study of Intraperitoneal Administration of Daptomycin in Peritoneal Infection
Acronym: DAPTODP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-005699-33
Record Dates: First submitted 2013-09-03; First posted 2013-12-04 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2017-01

CONDITIONS: Peritoneal Infection
Keywords: intraperitoneal; peritoneal dialysis; daptomycin; pharmacokinetics; peritonitis
MeSH Terms: conditions — Peritonitis

STUDY DESIGN:
Intervention Model Description: dose-finding study
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intraperitoneal daptomycin (Experimental): 3 first patients : 200mg/day 3 following patients : 300mg/day
  Interventions: Drug: intraperitoneal daptomycin

INTERVENTIONS:
Drug: intraperitoneal daptomycin — intraperitoneal daptomycin administartion and study of daptomycin kinetics

SUMMARY:
Peritoneal infection is still a frequent complication in peritoneal dialysis patients . In France, It contributes to the technique failure, responsible for about 20% of cases of transfer in hemodialysis. The risk of direct mortality is estimated at 1 to 6% according to studies. Peritoneal infection is involved in the dysfunction of the peritoneal membrane.

Based on the recommendations of the International Society for Peritoneal Dialysis, the intraperitoneal route is preferentially recommended. For many antibiotics, pharmacokinetics (intravenous and intraperitoneal) was studied and protocols for IP administration were validated.

Daptomycin, is a cyclic lipopeptide natural, active only on Gram-positive bacteria. It is presented as an alternative to vancomycin in infections resistant pathogens. The stability of daptomycin in peritoneal dialysis fluids (PDF) has been tested, and antimicrobial activity as well.

Seven patients were treated with daptomycin intraperitoneally successfully. But no study has reported pharmacokinetics of daptomycin via the IP route. We propose a pharmacokinetic study of daptomycin administered intraperitoneally in 12 patients on CAPD and with Gram-positive peritoneal infection.

DETAILED DESCRIPTION:
Methodology:

Prospective, open-label, non-randomized pharmacokinetic study. Daptomycin will be given IP in the CAPD fluid (200mg in 2L Nutrineal) once daily, in a 6 hours-dwell time. The process of dialysis is done four times per day : three during the day (6,6,and 4 h) and one time at night (8h). Duration of treatment depends on bacteria identified (14 or 21 days).

Analyses will be performed on data from all patients meeting the criteria for inclusion and exclusion.

For each patient, plasma, dialysate and urine kinetics will be studied.

For each parameter, mean and standard deviation are calculated.

Number of centers & patients:

One center, twelve patients.

Sample size justification:

This is an observational pharmacokinetic study of consecutive PD patients presenting to Caen University Hospital with peritoneal infection and who meet inclusion criterias over one year.

Population: CAPD patients with a Gram positive peritoneal infection

ELIGIBILITY:
Inclusion Criteria:

Patients > 18 years

* Hospitalized CAPD patients with Gram positive peritoneal infection : ISPD criterias
* Presence of two clinical signs and symptoms : abdominal pain, nausea, vomiting, diarrhea, fever and cloudy dialysate
* Peritoneal dialysate WBC>100/µL with at least 50% polymorphonuclear neutrophil cells
* Demonstration of bacteria on Gram stain or culture
* on peritoneal dialysis for at least 3 months
* written consent, obtained from either the patient, one of his/her relatives, the trusted person who was designated beforehand or, if not possible, emergency enrollment.
* patient has a life expectancy greater than 6 months

Exclusion Criteria:

* Known allergy to daptomycin
* Peritoneal infection with Gram negative only
* Patient with CPK>5UNL
* patients already treated with antibiotics, antifungals within 4 weeks prior to the event
* Patient with hepatic impairment
* Patient with arguments for an extra-peritoneal site of infection
* Patient with severe intercurrent illness (eg, hematologic malignancies, patients on chemotherapy)
* Infection by daptomycin-resistant germ
* HMGCoA reductase, fibrates or ciclosporin treatment
* Pregnant or breast-feeding women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 14 days
  Primary endpoint :
  Pharmacokinetics study : Evaluation of :
  * the maximum plasma concentration,
  * areas under the curve
  * compartments clearances,
  * the time during which dialysate concentration is greater than 20mg /L (5xEnterococcus CMI)

SECONDARY OUTCOMES:
tolerance | 14 days
  CPK<5N

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Lobbedez, Pr, Principal Investigator — University Hospital, Caen; Maxence FICHEUX, Dr, Study Director — University Hospital, Caen
Locations (1):
- Néphrologie CHU de Caen, Caen, France